CLINICAL TRIAL: NCT00124046
Title: Treatment of Persistent Urinary Incontinence in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H05-70276
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence in Children; Surgical Section of the Filum Terminale; Occult Tethered Cord Syndrome; Urodynamic Scale; Enuresis-Specific Quality of Life Scale
MeSH Terms: conditions — Urinary Incontinence | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical (Active Comparator)
  Interventions: Procedure: Surgery
- Medical Treatment (Active Comparator)
  Interventions: Procedure: Medical Treatment

INTERVENTIONS:
Procedure: Surgery — Surgery for this diagnosis is a standard of care, as is the medical treatment. We are comparing the two
  Arms: Surgical
Procedure: Medical Treatment — Surgery for this diagnosis is a standard of care, as is the medical treatment. We are comparing the two
  Arms: Medical Treatment

SUMMARY:
The purpose of this study is to determine whether surgical section of the filum terminale in children, when added to standard medical therapy, will result in a reliable and clinically-significant improvement in two main markers of incontinence within/at 12 months after treatment.

DETAILED DESCRIPTION:
Eight % to sixteen % of school-aged children or approximately 50,000 children in British Columbia (BC) suffer from persistent urinary incontinence (i.e., beyond age 5 years, when continence is usually achieved). Prevalence decreases with age, yet studies indicate that 10%-25% of healthy adolescents and young adults also suffer from incontinence. Persistent incontinence has profound social, emotional and behavioral impacts, and adversely affects the quality of life of affected children and their families.

Typical management of incontinence in these patients includes repeated visits to the family doctor and long-term lifestyle changes and/or prescription use. Each year in BC, family doctors refer about 4500 children to pediatric urologists at BC Children's Hospital (BCCH). BCCH is the only tertiary care facility for children and youth in the province, so that children and parents come from all over BC for these appointments and for diagnostic urodynamics testing. Of these children who are evaluated by pediatric urologists each year, approximately 900 (20%) are designated as having dysfunctional voiding. In this group, following one year of non-responsiveness to medical treatment (medication, lifestyle), the urologist may refer the child to neurosurgery for assessment and possible surgery.

In recent years, the referral rate of children with incontinence to BCCH Neurosurgery has increased markedly from 1-2 to 12-15 children per year. This referral is because urinary incontinence in children is one of the clinical features of a tethered cord syndrome. In this syndrome, the lower end of the spinal cord (the conus) is pulled down lower than normal by a thickened band of tissue called the filum terminale, which runs inferiorly from the bottom of the spinal cord. This "tethered" condition can be treated by surgical section of the filum terminale. More recently, the concept of an occult tethered cord syndrome (OTCS) has been proposed; in OTCS, clinical symptoms (e.g., incontinence) are consistent with a tethered cord syndrome, but the conus ends at a normal location. The concept of the OTCS is controversial, and it is not yet clear whether or not section of the filum is appropriate. Filum section is a relatively minor procedure (akin to appendectomy) that requires general anesthesia during day surgery. In uncontrolled case series, section of the filum terminale in children with OTCS resulted in a 60%-97% improvement in symptoms.

Given this evidence that section of the filum may improve incontinence symptoms, urologists are keen to refer more patients to neurosurgeons. Furthermore, families are demanding more tests and options, and are ready to pursue surgery as treatment of their child's incontinence. This suggests that the referral rate to Neurosurgery will continue to increase, and there will be a crucial requirement to develop standard policies and procedures related to offering this surgery to children with incontinence. As yet, however, the effectiveness and appropriateness of the surgery have not been evaluated systematically.

To investigate this matter a comparison will be made between two randomized groups. One group will undergo early tethered cord release by section of the filum terminale through a limited posterior lumbar spinal exposure and continued medical therapy for 12 months. This group will be compared to a second that has continued standard medical therapy without surgical intervention for a further 12 months. This comparison will be made based on physiological markers of urinary incontinence, as measured by a urodynamic scale; and quality of life, as measured by a validated enuresis-specific quality of life scale. The intervention will be considered to be successful if it improves the urodynamic score by 20%, and the quality of life of the child and his family are significantly improved.

ELIGIBILITY:
Inclusion Criteria:

Urologic Inclusion Criteria:

* Primary or secondary daytime urinary incontinence, persistent over 12 months of medical treatment
* An abnormal 3 day voiding diary compiled over a 3 week voiding period completed after 12 months of medical treatment
* Normal bladder ultrasound (if bladder ultrasound shows more than minimal bladder thickening [>3.0mm at 50% filling of expected capacity or less] then a voiding cystourethrogram [VCUG] will be required to rule out bladder outlet obstruction)
* Abnormal urodynamic testing

Radiologic Inclusion Criteria:

* Normal position conus medullaris
* Any size filum terminale
* Any amount of fat in the filum terminale
* Terminal syringomyelia of less than one bony level is acceptable
* Lumbar bifid spinal lamina is acceptable

Exclusion Criteria:

* Patients with evidence of significant, progressive, lower extremity motor or sensory deficits, with evidence of progression over the previous 6 months
* The presence of cutaneous markings on the back, in the absence of confirmatory magnetic resonance imaging (MRI) findings of a specific spinal dysraphism does not exclude the patient from participation

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2005-09; Primary Completion 2014-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Quality of life, as measured by a validated enuresis-specific quality of life scale

SECONDARY OUTCOMES:
Any of the following radiographic findings leads to improved response to section of the filum: fat in the filum terminale, thickened filum terminale, presence of bifid lamina
Presence of a growth spurt in the 6 months following the section of the filum compared to the 6 months prior
Duration of urinary symptoms is negatively associated with improvement in urinary function
The following subtle neurological abnormalities are predictors of good outcome following filum section: strength or sensory dysfunction, clinical symptoms of back or leg pain, inability to touch toes with forward flexion
Section of the filum terminale leads to reduced frequency of urinary infections in the 12 months following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Paul Steinbok, MB, BS, FRCSC, Principal Investigator — Children's and Women's Health Centre of British Columbia
Locations (1):
- Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Steinbok P, MacNeily AE, Hengel AR, Afshar K, Landgraf JM, Hader W, Pugh J. Filum Section for Urinary Incontinence in Children with Occult Tethered Cord Syndrome: A Randomized, Controlled Pilot Study. J Urol. 2016 Apr;195(4 Pt 2):1183-8. doi: 10.1016/j.juro.2015.09.082. Epub 2016 Feb 28. PMID 26926544